CLINICAL TRIAL: NCT06612502
Title: The Effect of Percussion Massage Therapy on the Recovery of Delayed Onset Muscle Soreness in Physically Active Young Men
Brief Title: The Effect of Percussion Massage Therapy on the Recovery of DOMS in Physically Active Young Men Delayed Onset Muscle Soreness = DOMS
Acronym: Required
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanxi Normal University (Other)
Responsible Party: Principal Investigator, Haiwei Li, Professor, Shanxi Normal University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-0803
Record Dates: First submitted 2024-09-21; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-05

CONDITIONS: Delayed Onset Muscle Soreness (DOMS)
Keywords: Delayed Onset Muscle Soreness; Percussion massage therapy; Stretching; Recovery
MeSH Terms: interventions — Muscle Stretching Exercises

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Static Stretching group (Active Comparator): The static stretching protocol comprised eight exercises, performed for 30 seconds per bilateral muscle group (with the exception of the sitting toe touch and butterfly stretch), and included the hip, knee, and ankle. Each subject completed each stretch before progressing to the subsequent one. The stretches were maintained until the subject experienced mild discomfort, but not pain.
  Interventions: Behavioral: Static stretching
- short-time PMT group (Experimental): The PMT was performed by the two physiotherapists using an OUTSO 06® Fascia Gun equipped with a 5 cm diameter soft attachment head. Throughout the PMT, the physiotherapists carefully maintained a consistent level of moderate pressure on the skin, and followed the direction of the muscle fibers. In the S-PMT group, the treatment was applied for 25minutes.
  Interventions: Device: Fascia gun ( Short-time PMT )
- long-time PMT group (Experimental): The PMT was performed by the two physiotherapists using an OUTSO 06® Fascia Gun equipped with a 5 cm diameter soft attachment head. Throughout the PMT, the physiotherapists carefully maintained a consistent level of moderate pressure on the skin, and followed the direction of the muscle fibers. In the L-PMT group, the treatment was applied for 40 minutes.
  Interventions: Device: Fascia gun ( Long-time PMT )

INTERVENTIONS:
Behavioral: Static stretching — The static stretching protocol comprised eight exercises, performed for 30 seconds per bilateral muscle group (with the exception of the sitting toe touch and butterfly stretch), and included the hip, knee, and ankle. The subjects were instructed to perform the following sequence of stretches: forward lunge, supine knee flexion, lateral quadriceps stretch, sitting toe touch, semi-straddle, straddle, butterfly stretch, and a straight knee ankle extensor wall stretch. Each subject completed each stretch before progressing to the subsequent one. The stretches were maintained until the subject experienced mild discomfort, but not pain.
  Arms: Static Stretching group
Device: Fascia gun ( Short-time PMT ) — The PMT was performed by the two physiotherapists using an OUTSO 06® Fascia Gun equipped with a 5 cm diameter soft attachment head and the vibration frequency was 53 Hz. The targeted muscles included the quadriceps, adductors, hamstrings, iliotibial band, and gluteal muscles for both sides. Throughout the PMT, the physiotherapists carefully maintained a consistent level of moderate pressure on the skin, and followed the direction of the muscle fibers. The short time PMT was applied for 2.5 minutes per muscle site for a total of 25 minutes.
  Arms: short-time PMT group
Device: Fascia gun ( Long-time PMT ) — The PMT was performed by the two physiotherapists using an OUTSO 06® Fascia Gun equipped with a 5 cm diameter soft attachment head and the vibration frequency was 53 Hz. The targeted muscles included the quadriceps, adductors, hamstrings, iliotibial band, and gluteal muscles for both sides. Throughout the PMT, the physiotherapists carefully maintained a consistent level of moderate pressure on the skin, and followed the direction of the muscle fibers. The long time PMT was applied for 4 minutes per muscle site for a total of 40 minutes.
  Arms: long-time PMT group

SUMMARY:
The goal of this clinical trial is to learn the effect of percussion massage therapy (PMT) on the recovery of delayed onset muscle soreness (DOMS) in physically active young men.

The main question it aims to answer is:

Compared with static stretching, Do 25 minutes and 40 minutes of PMT can decrease pain and increase the rang of motion of knee of low limb DOMS in physically active young men? Compared with static stretching, Do 25 minutes and 40 minutes of PMT sessions can increase power and improve the neuromuscular electrophysiology of low limb DOMS in physically active young men?

Researchers will compare 25 minutes and 40 minutes of PMT to a static stretching to see if different times of PMT are better to treat DOMS.

Participants will： Undergo squats to induce low limb DOMS. Receive static stretching, 25 minutes and 40 minutes of PMT, respectively for three times.

Visit the lab for four times in one week for tests.

ELIGIBILITY:
Inclusion Criteria:

Regularly participate in physical activity, have no contraindications to exercise, and volunteered to participate in this study

Exclusion Criteria:

Participants consumed alcohol and exercised vigorously throughout the formal experiment or they underwent interventions other than those planned for the experiment.

Ages: 19 Years to 23 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-21 (Actual)

PRIMARY OUTCOMES:
Muscle pain | From enrollment to the end of treatment for 3 days
  The intensity of muscle pain was quantified using the visual analogue scale (VAS), which comprises a 10-cm straight line with one end labelled (score of 0) and the other end labelled intolerable pain (score of 10). Subjects were required to provide a rating of their perceived lower-limb muscle soreness for each leg on a scale of one (no soreness) to ten (maximal soreness). Two measurements were recorded on the VAS scale, and the average was calculated.
Knee joint ROM | From enrollment to the end of treatment for 3 days
  A modified kneeling lunge was employed to assess knee joint ROM. The procedure was as follows: the subjects left leg was bent at the knee, the thigh was parallel to the ground, and the left lower leg was perpendicular to the ground; the right leg was bent at the knee, and the upper body was maintained in an upright position. The subject was required to adjust the position in order to stretch the right hip to the point of discomfort. The angle to which the right hip was stretched was measured and used as a criterion for subsequent measurement of the ROM. The investigator then bent the subjects right knee until the level of discomfort was reached. At this point, the angle between the thigh and calf was recorded using a goniometer, with the following landmarks: the lateral malleolus, the lateral epicondyle, and the center of the vastus lateralis. A larger angle indicated a smaller ROM of the knee joint.
CMJ | From enrollment to the end of treatment for 3 days
  The CMJ was performed in accordance with the established methodology described in the existing literature, and the variables with the CMJ were evaluated using a BTS P-6000 three-dimensional force platform (BTS Bioengineering, Milan, Italy), with a sampling frequency of 1000 Hz. Three trials were conducted for each subject, and the highest vertical jump height was selected for analysis. The variables obtained included the jump height, the peak ground reaction force during the propulsion phase, and the propulsion impulse. The jump height was calculated from the time spent in the air. The peak ground reaction force was obtained from the force-time curve, and the calculation of the propulsion impulse was based on the previous literature.
Surface EMG | From enrollment to the end of treatment for 3 days
  In this study, wireless sEMG (Noraxon USA Inc., Scottsdale, AZ, USA) was employed to collect the integrated EMG (iEMG) from the vastus medialis, rectus femoris, and vastus lateralis during the completion of the CMJ on the dominant leg, with a sampling frequency of 1000 Hz. The skin surface was prepared by abrasion and alcohol swabs. Disposable Ag-AgCl circular surface electrodes (4 mm diameter) were filled with electrode jelly and attached 2.5 cm apart to each muscle. Once the EMG test was complete, the raw data were processed using Noraxon TeleMyo (Noraxon USA Inc., Scottsdale,AZ, USA) software for rectification, smoothing, and filtering. In order to eliminate the effect of time phase, the signal was partitioned in 10-ms windows to find for each muscle and each subject its maximal activation over CMJ (iEMGmax). iEMGmax was considered to be 100%. Then, the iEMG of CMJ duration was divided by the time (iEMG/T) and expressed in percentage iEMGmax.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanxi Normal University, Taiyuan, Shanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li H, Luo L, Zhang J, Cheng P, Wu Q, Wen X. The effect of percussion massage therapy on the recovery of delayed onset muscle soreness in physically active young men-a randomized controlled trial. Front Public Health. 2025 Mar 26;13:1561970. doi: 10.3389/fpubh.2025.1561970. eCollection 2025. PMID 40206177